CLINICAL TRIAL: NCT00344279
Title: Changes in HIV Viral Load in Patients Undergoing Treatment for Filarial Infection
Brief Title: Changes in HIV Viral Load in Patients Undergoing Treatment for Filariasis
Status: Completed | Type: Observational
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 999905220; 05-I-N220
Record Dates: First submitted 2006-06-23; First posted 2006-06-26 (Estimated); Last update posted 2017-07-02 (Actual); Status verified 2012-01-31

CONDITIONS: Filarial Infection; HIV Infections
Keywords: Coinfection; AIDS; Lymphatic Filariasis; Diethylcarbamazine (DEC); Albendazole
MeSH Terms: conditions — HIV Infections; Coinfection; Acquired Immunodeficiency Syndrome; Elephantiasis, Filarial

SUMMARY:
This study, sponsored by the National Institutes of Health and the Tuberculosis Research Centre and YRG-Care in Chennai, India, will examine how treatment of lymphatic filariasis in HIV-infected patients influences the amount of HIV virus in the blood and the progression of HIV infection to AIDS. Filarial infections are common in Chennai, and it is important to understand whether treatment of filariasis affects the course of HIV disease. The information gained from this study could be used to modify treatments for people both with HIV and filarial infections.

Patients 18 years of age and older who are receiving treatment for HIV infection at the Government Hospital HIV clinic or YRG-Care may be eligible for this study. Two groups of patients will be recruited - patients with both HIV and filarial infections, and patients who have HIV infection alone, without filariasis. Candidates are screened with a medical history and review of medical records, physical examination, and blood and stool tests. Women have a urine pregnancy test.

Within one month of screening, all participants receive a single dose of diethylcarbamazine and albendazole, a drug regimen commonly used to treat filarial infection. Patients are followed closely for the first 2 weeks after treatment to check for side effects. They are then seen at 1, 3, 6 and 12 months after the treatment dose for a physical examination and blood test.

DETAILED DESCRIPTION:
To determine the effect of pre-existing filarial infection and its treatment on viral burden and clinical parameters in patients infected with HIV, this study aims to follow plasma HIV loads, CD4 counts, and clinical parameters in a population of HIV-infected individuals co-infected with Wuchereria bancrofti, prior to and after treatment of filarial infection. The study individuals will be drawn from the patient cohort followed by the HIV Clinic at the Government General Hospital and the Tuberculosis Research Centre, Chennai, India, or those from YRG-Care (Chennai, India), an area endemic for lymphatic filariasis (LF) and where the prevalence of HIV infection in the general population is about 7%. These patients are adults of all ages, both males and females, come from the states of Tamil Nadu and Andhra Pradhesh. Having established as part of a previous protocol (01-I-N022) an HIV/filarial coprevalence of 6-10% based on W. bancrofti circulating antigen detection in HIV-positive and -negative individuals, patients in whom co-infection with HIV and LF has been diagnosed will be paired with two HIV-positive (but filarial antigen negative) clinic controls matched for age, gender, viral load antiretroviral therapy and CD4 count. All efforts will be made to connect study participants with programs for antiretroviral distribution. Within a month of a baseline clinical evaluation, patients and controls will receive a single dose of the combination of diethylcarbamazine/albendazole (the drug combination given as part of national campaigns to eliminate LF) and will then be followed with viral loads, CD4 counts and clinical examinations at one week, as well as 1, 3, 6 and 12 months after the administration. By assessing these changes, the influence of a co-existing filarial infection on plasma HIV viral load, CD4 count and clinical course can be determined. At the end of the study period, all participants will be re-assessed for filarial antibody and antigen to ensure absence of the parasite. Any patient who has evidence of ongoing filarial infection with W. bancrofti will be re-treated with DEC/albendazole.

ELIGIBILITY:
* INCLUSION CRITERIA:

Greater than 18 years of age.

Ability to give informed consent

HIV positive

If on antiretrovirals or treatment for opportunistic infections, have it be a stable maintenance period of at least 2 months

Male or female, providing women are neither pregnant nor breast-feeding

Willingness to adhere to the testing schedule of the protocol and to provide small amounts of blood (5 ml) on multiple occasions

Willingness to be treated with DEC/albendazole

Willingness, if female, to be tested for pregnancy and to be informed of the test result

Willingness to have samples stored for future research

EXCLUSION CRITERIA:

Acutely ill at the time of enrollment into the study i.e. newly diagnosed with an opportunistic infection and not yet stabilized on a treatment regime.

Hemoglobin less than 9 g/l for women and less than 10 g/l for men

AST, ALT greater than 5 times normal

Evidence of acute HIV infection (acute antiretroviral syndrome)

Active tuberculosis or known tuberculosis

A true allergy to DEC or albendazole

At the discretion of the investigator if it is felt that someone is not appropriate for the study (i.e. known active drug use, patient with history of chronic noncompliance in clinic visits)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1000 (Estimated)
Dates: Start 2005-08-08; Study Completion 2012-01-31

CONTACTS AND LOCATIONS:
Locations (3):
- India (3):
  - Government General Hospital, Chennai
  - Tuberculosis Research Centre, Chennai
  - YRG Care, Chennai

REFERENCES:
- [Background] Bloland PB, Wirima JJ, Steketee RW, Chilima B, Hightower A, Breman JG. Maternal HIV infection and infant mortality in Malawi: evidence for increased mortality due to placental malaria infection. AIDS. 1995 Jul;9(7):721-6. doi: 10.1097/00002030-199507000-00009. PMID 7546417
- [Background] Brown M, Kizza M, Watera C, Quigley MA, Rowland S, Hughes P, Whitworth JA, Elliott AM. Helminth infection is not associated with faster progression of HIV disease in coinfected adults in Uganda. J Infect Dis. 2004 Nov 15;190(10):1869-79. doi: 10.1086/425042. Epub 2004 Oct 20. PMID 15499545
- [Background] Bush CE, Donovan RM, Markowitz NP, Kvale P, Saravolatz LD. A study of HIV RNA viral load in AIDS patients with bacterial pneumonia. J Acquir Immune Defic Syndr Hum Retrovirol. 1996 Sep;13(1):23-6. doi: 10.1097/00042560-199609000-00004. PMID 8797682
- [Derived] Talaat KR, Babu S, Menon P, Kumarasamy N, Sharma J, Arumugam J, Dhakshinamurthy K, Srinivasan R, Poongulali S, Gu W, Fay MP, Swaminathan S, Nutman TB. Treatment of W. bancrofti (Wb) in HIV/Wb coinfections in South India. PLoS Negl Trop Dis. 2015 Mar 20;9(3):e0003622. doi: 10.1371/journal.pntd.0003622. eCollection 2015 Mar. PMID 25793933